CLINICAL TRIAL: NCT05201521
Title: The Chinese Functional Movement Disorders Registry Study
Brief Title: Chinese FMDs Registry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SN-01
Record Dates: First submitted 2021-12-23; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Functional Movement Disorders
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Chinese Functional Movement Disorders Registry (FMDs-China) is to develop a database of patients with Functional Movement Disorders (FMDs) in China.

DETAILED DESCRIPTION:
Functional movement disorders (FMDs), also known as psychogenic movement disorders (PMDs), formerly known as "hysteria or hysteria", is a representative functional nervous system disease. It has been reported in Europe and America that FMDs patients account for 3% - 6% of all patients in the outpatient department of motor disorders, but there is no relevant data report in China so far. From the current research, the incidence rate has gradually increased significantly. However, the research about the pathogenesis and diagnosis of such diseases is rare. These studies have the problem of small sample size and still lack large randomized controlled studies to demonstrate the long-term efficacy of different treatments. And in China, there are nearly no reliable research and the lack of basic understanding makes it a "gray area" for the diagnosis and treatment of FMDs.

The purpose of this observational study is to prospectively register the information of patients with FMDs nationwide, establishing a Chinese multicenter FMDs China cohort; understanding the demographic characteristics, clinical characteristics and symptom characteristics, neuropsychological test, electrophysiological and imaging characteristics, drug use, etc. what's more, it lays a foundation for the research on the etiology and treatment in the second stage of this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Age 18-80;
* Patients clinically diagnosed with functional movement disorders according to the Fahn-Williams criteria;
* Patients who are willing to provide information such as disease history and cooperate with physical examination and examination;

Exclusion Criteria:

* Patients with definite organic dyskinesia;
* There are other causes of dyskinesia such as fatigue, pain, hyperthyroidism, chronic alcoholism, and drug use;
* Those who suffer from serious physical diseases and are unable to cooperate;
* Those who do not cooperate or refuse to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 100 patents coming from hospitals or communities in mainland China
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-27 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-01-27 (Estimated)

PRIMARY OUTCOMES:
The symptom characteristics | baseline
  Symptom characteristics such as tremor, type of dystonia, Parkinson's like symptoms, myoclonus, etc.
The symptom characteristics | 0.5 years
  Symptom characteristics such as tremor, type of dystonia, Parkinson's like symptoms, myoclonus, etc.
The symptom characteristics | 1.5 years
  Symptom characteristics such as tremor, type of dystonia, Parkinson's like symptoms, myoclonus, etc.
The symptom characteristics | 2 years
  Symptom characteristics such as tremor, type of dystonia, Parkinson's like symptoms, myoclonus, etc.
The movement disorder attack video | baseline
  The video is taken as the protocol below: full body view of the participant sitting in a chair with arm rests (15 seconds); close up of face and neck (15 seconds), the participant was then asked to recite the months of the year; full body view sitting with hands supine resting on thighs (15 seconds); arms extended at shoulder height with hands in pronation (10 seconds); ﬁnger-nose test (5 repetitions); thumb and index-finger finger taps (15 seconds); heel taps (15 seconds); moving from sitting to standing; standing with posture uncorrected (10 seconds); standing with feet touching (10 seconds); and ﬁnally walking 5 meters, turn and walking back to the starting position (using aids if necessary). All video was ﬁlmed in a frontal view.
The movement disorder attack video | 0.5 years
  The video is taken as the protocol below: full body view of the participant sitting in a chair with arm rests (15 seconds); close up of face and neck (15 seconds), the participant was then asked to recite the months of the year; full body view sitting with hands supine resting on thighs (15 seconds); arms extended at shoulder height with hands in pronation (10 seconds); ﬁnger-nose test (5 repetitions); thumb and index-finger finger taps (15 seconds); heel taps (15 seconds); moving from sitting to standing; standing with posture uncorrected (10 seconds); standing with feet touching (10 seconds); and ﬁnally walking 5 meters, turn and walking back to the starting position (using aids if necessary). All video was ﬁlmed in a frontal view.
The movement disorder attack video | 1.5 years
  The video is taken as the protocol below: full body view of the participant sitting in a chair with arm rests (15 seconds); close up of face and neck (15 seconds), the participant was then asked to recite the months of the year; full body view sitting with hands supine resting on thighs (15 seconds); arms extended at shoulder height with hands in pronation (10 seconds); ﬁnger-nose test (5 repetitions); thumb and index-finger finger taps (15 seconds); heel taps (15 seconds); moving from sitting to standing; standing with posture uncorrected (10 seconds); standing with feet touching (10 seconds); and ﬁnally walking 5 meters, turn and walking back to the starting position (using aids if necessary). All video was ﬁlmed in a frontal view.
The movement disorder attack video | 2 years
  The video is taken as the protocol below: full body view of the participant sitting in a chair with arm rests (15 seconds); close up of face and neck (15 seconds), the participant was then asked to recite the months of the year; full body view sitting with hands supine resting on thighs (15 seconds); arms extended at shoulder height with hands in pronation (10 seconds); ﬁnger-nose test (5 repetitions); thumb and index-finger finger taps (15 seconds); heel taps (15 seconds); moving from sitting to standing; standing with posture uncorrected (10 seconds); standing with feet touching (10 seconds); and ﬁnally walking 5 meters, turn and walking back to the starting position (using aids if necessary). All video was ﬁlmed in a frontal view.
The Simplified Functional Movement Disorders Rating Scale | baseline
  The Simplified Functional Movement Disorders Rating Scale (S-FMDRS) is used to estimate the provide a snapshot symptom severity score and provide information on phenomenology, anatomical distribution, duration, and functional impact of abnormal movement. Symptom severity at 7 body region and 2 functions (gait and speech) are rated from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe). A duration score was assigned to each body region and function (estimated amount of time in the video during which symptoms are observed at the body region), rated from 0 to 3 (0 = none; 1 = symptomatic movement spotted at least once or only a few times; 2 = symptom is intermittent but frequent so that there are periods during which it is absent or does not affect purposeful movement; 3 = the symptom is evident continuously). The total score is 54, the minimum is 0, higher scores indicate more severe disease.
The Simplified Functional Movement Disorders Rating Scale | 0.5 years
  The Simplified Functional Movement Disorders Rating Scale (S-FMDRS) is used to estimate the provide a snapshot symptom severity score and provide information on phenomenology, anatomical distribution, duration, and functional impact of abnormal movement. Symptom severity at 7 body region and 2 functions (gait and speech) are rated from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe). A duration score was assigned to each body region and function (estimated amount of time in the video during which symptoms are observed at the body region), rated from 0 to 3 (0 = none; 1 = symptomatic movement spotted at least once or only a few times; 2 = symptom is intermittent but frequent so that there are periods during which it is absent or does not affect purposeful movement; 3 = the symptom is evident continuously). The total score is 54, the minimum is 0, higher scores indicate more severe disease.
The Simplified Functional Movement Disorders Rating Scale | 1 years
  The Simplified Functional Movement Disorders Rating Scale (S-FMDRS) is used to estimate the provide a snapshot symptom severity score and provide information on phenomenology, anatomical distribution, duration, and functional impact of abnormal movement. Symptom severity at 7 body region and 2 functions (gait and speech) are rated from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe). A duration score was assigned to each body region and function (estimated amount of time in the video during which symptoms are observed at the body region), rated from 0 to 3 (0 = none; 1 = symptomatic movement spotted at least once or only a few times; 2 = symptom is intermittent but frequent so that there are periods during which it is absent or does not affect purposeful movement; 3 = the symptom is evident continuously). The total score is 54, the minimum is 0, higher scores indicate more severe disease.
The Simplified Functional Movement Disorders Rating Scale | 1.5 years
  The Simplified Functional Movement Disorders Rating Scale (S-FMDRS) is used to estimate the provide a snapshot symptom severity score and provide information on phenomenology, anatomical distribution, duration, and functional impact of abnormal movement. A duration score was assigned to each body region and function (estimated amount of time in the video during which symptoms are observed at the body region), rated from 0 to 3 (0 = none; 1 = symptomatic movement spotted at least once or only a few times; 2 = symptom is intermittent but frequent so that there are periods during which it is absent or does not affect purposeful movement; 3 = the symptom is evident continuously). The total score is 54, the minimum is 0, higher scores indicate more severe disease.
The Simplified Functional Movement Disorders Rating Scale | 2 years
  The Simplified Functional Movement Disorders Rating Scale (S-FMDRS) is used to estimate the provide a snapshot symptom severity score and provide information on phenomenology, anatomical distribution, duration, and functional impact of abnormal movement. A duration score was assigned to each body region and function (estimated amount of time in the video during which symptoms are observed at the body region), rated from 0 to 3 (0 = none; 1 = symptomatic movement spotted at least once or only a few times; 2 = symptom is intermittent but frequent so that there are periods during which it is absent or does not affect purposeful movement; 3 = the symptom is evident continuously). The total score is 54, the minimum is 0, higher scores indicate more severe disease.

SECONDARY OUTCOMES:
Hamilton Depression Scale | baseline
  Hamilton Depression Scale (HAMD) was designed to measure frequency and intensity of depressive symptoms in individuals with major depressive disorder. Scores between 0 and 6 do not indicate the presence of depression' scores between 7 and 17 indicate mild depression' scores between 18 and 24 indicate moderate depression' and scores over 24 indicate severe depression.
Hamilton Depression Scale | 0.5 years
  Hamilton Depression Scale (HAMD) was designed to measure frequency and intensity of depressive symptoms in individuals with major depressive disorder. Scores between 0 and 6 do not indicate the presence of depression' scores between 7 and 17 indicate mild depression' scores between 18 and 24 indicate moderate depression' and scores over 24 indicate severe depression.
Hamilton Depression Scale | 1 years
  Hamilton Depression Scale (HAMD) was designed to measure frequency and intensity of depressive symptoms in individuals with major depressive disorder. Scores between 0 and 6 do not indicate the presence of depression' scores between 7 and 17 indicate mild depression' scores between 18 and 24 indicate moderate depression' and scores over 24 indicate severe depression.
Hamilton Depression Scale | 1.5 years
  Hamilton Depression Scale (HAMD) was designed to measure frequency and intensity of depressive symptoms in individuals with major depressive disorder. Scores between 0 and 6 do not indicate the presence of depression' scores between 7 and 17 indicate mild depression' scores between 18 and 24 indicate moderate depression' and scores over 24 indicate severe depression.
Hamilton Depression Scale | 2 years
  Hamilton Depression Scale (HAMD) was designed to measure frequency and intensity of depressive symptoms in individuals with major depressive disorder. Scores between 0 and 6 do not indicate the presence of depression' scores between 7 and 17 indicate mild depression' scores between 18 and 24 indicate moderate depression' and scores over 24 indicate severe depression.
Beck Anxiety Inventory | baseline
  Beck Anxiety Inventory (BAI) is a self-report measure of anxiety.The total score is calculated by finding the sum of the 21 items.Score of 0 - 21 = low anxiety;Score of 22 - 35 = moderate anxiety;Score of 36 and above = potentially concerning levels of anxiety
Beck Anxiety Inventory | 0.5 years
  Beck Anxiety Inventory (BAI) is a self-report measure of anxiety.The total score is calculated by finding the sum of the 21 items.Score of 0 - 21 = low anxiety;Score of 22 - 35 = moderate anxiety;Score of 36 and above = potentially concerning levels of anxiety
Beck Anxiety Inventory | 1 years
  Beck Anxiety Inventory (BAI) is a self-report measure of anxiety.The total score is calculated by finding the sum of the 21 items.Score of 0 - 21 = low anxiety;Score of 22 - 35 = moderate anxiety;Score of 36 and above = potentially concerning levels of anxiety
Beck Anxiety Inventory | 1.5 years
  Beck Anxiety Inventory (BAI) is a self-report measure of anxiety.The total score is calculated by finding the sum of the 21 items.Score of 0 - 21 = low anxiety;Score of 22 - 35 = moderate anxiety;Score of 36 and above = potentially concerning levels of anxiety
Beck Anxiety Inventory | 2 years
  Beck Anxiety Inventory (BAI) is a self-report measure of anxiety.The total score is calculated by finding the sum of the 21 items.Score of 0 - 21 = low anxiety;Score of 22 - 35 = moderate anxiety;Score of 36 and above = potentially concerning levels of anxiety
symptom check list-90 | baseline
  symptom check list-90 (SLC-90) is a 90-item self-report symptom inventory to measure psychological symptoms and psychological distress including Somatization, Obsessive-Compulsive, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, and Psychoticism. Positive items refer to items with a single item score ≥ 2. According to the China national norm results, if the total score exceeds 160 points, or the number of positive items exceeds 43, the screening should be considered positive and further examination is required. The score of the total symptom index is between 1 and 1.5, indicating that the subject feels no symptoms; between 1.5 and 2.5, it indicates that the subject feels a little symptom, but it occurs infrequently; between 2.5 and 3.5, the severity was mild to moderate; between 3.5 and 4.5, the severity was moderate to severe; between 4.5 and 5, the frequency and intensity of symptoms are severe.
symptom check list-90 | 0.5 years
  symptom check list-90 (SLC-90) is a 90-item self-report symptom inventory to measure psychological symptoms and psychological distress including Somatization, Obsessive-Compulsive, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, and Psychoticism. Positive items refer to items with a single item score ≥ 2. According to the China national norm results, if the total score exceeds 160 points, or the number of positive items exceeds 43, the screening should be considered positive and further examination is required. The score of the total symptom index is between 1 and 1.5, indicating that the subject feels no symptoms; between 1.5 and 2.5, it indicates that the subject feels a little symptom, but it occurs infrequently; between 2.5 and 3.5, the severity was mild to moderate; between 3.5 and 4.5, the severity was moderate to severe; between 4.5 and 5, the frequency and intensity of symptoms are severe.
symptom check list-90 | 1 years
  symptom check list-90 (SLC-90) is a 90-item self-report symptom inventory to measure psychological symptoms and psychological distress including Somatization, Obsessive-Compulsive, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, and Psychoticism. Positive items refer to items with a single item score ≥ 2. According to the China national norm results, if the total score exceeds 160 points, or the number of positive items exceeds 43, the screening should be considered positive and further examination is required. The score of the total symptom index is between 1 and 1.5, indicating that the subject feels no symptoms; between 1.5 and 2.5, it indicates that the subject feels a little symptom, but it occurs infrequently; between 2.5 and 3.5, the severity was mild to moderate; between 3.5 and 4.5, the severity was moderate to severe; between 4.5 and 5, the frequency and intensity of symptoms are severe.
symptom check list-90 | 1.5 years
  symptom check list-90 (SLC-90) is a 90-item self-report symptom inventory to measure psychological symptoms and psychological distress including Somatization, Obsessive-Compulsive, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, and Psychoticism. Positive items refer to items with a single item score ≥ 2. According to the China national norm results, if the total score exceeds 160 points, or the number of positive items exceeds 43, the screening should be considered positive and further examination is required. The score of the total symptom index is between 1 and 1.5, indicating that the subject feels no symptoms; between 1.5 and 2.5, it indicates that the subject feels a little symptom, but it occurs infrequently; between 2.5 and 3.5, the severity was mild to moderate; between 3.5 and 4.5, the severity was moderate to severe; between 4.5 and 5, the frequency and intensity of symptoms are severe.
symptom check list-90 | 2 years
  symptom check list-90 (SLC-90) is a 90-item self-report symptom inventory to measure psychological symptoms and psychological distress including Somatization, Obsessive-Compulsive, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, and Psychoticism. Positive items refer to items with a single item score ≥ 2. According to the China national norm results, if the total score exceeds 160 points, or the number of positive items exceeds 43, the screening should be considered positive and further examination is required. The score of the total symptom index is between 1 and 1.5, indicating that the subject feels no symptoms; between 1.5 and 2.5, it indicates that the subject feels a little symptom, but it occurs infrequently; between 2.5 and 3.5, the severity was mild to moderate; between 3.5 and 4.5, the severity was moderate to severe; between 4.5 and 5, the frequency and intensity of symptoms are severe.
clinical global impression severity scale | baseline
  clinical global impression severity scale (CGI-S) is used to estimate the overall measure of severity of a patient's illness. CGI-S (categories: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = extremely ill
clinical global impression severity scale | 0.5 years
  clinical global impression severity scale (CGI-S) is used to estimate the overall measure of severity of a patient's illness. CGI-S (categories: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = extremely ill
clinical global impression severity scale | 1 years
  clinical global impression severity scale (CGI-S) is used to estimate the overall measure of severity of a patient's illness. CGI-S (categories: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = extremely ill
clinical global impression severity scale | 1.5 years
  clinical global impression severity scale (CGI-S) is used to estimate the overall measure of severity of a patient's illness. CGI-S (categories: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = extremely ill
clinical global impression severity scale | 2 years
  clinical global impression severity scale (CGI-S) is used to estimate the overall measure of severity of a patient's illness. CGI-S (categories: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = extremely ill
Clinical global improvement scale | baseline
  Clinical Global Impression Scale-improvement scale (CGI-I) has been widely utilized as an efficacy measure in clinical drug trials in different mental disorders.0: Very much; 1: improved; 2: Much improved; 3: Minimally improved; 4: No change; 5: Minimally worse; 6: Much worse; 7: Very much worse
Clinical global improvement scale | 0.5 years
  Clinical Global Impression Scale-improvement scale (CGI-I) has been widely utilized as an efficacy measure in clinical drug trials in different mental disorders.0: Very much; 1: improved; 2: Much improved; 3: Minimally improved; 4: No change; 5: Minimally worse; 6: Much worse; 7: Very much worse
Clinical global improvement scale | 1 year
  Clinical Global Impression Scale-improvement scale (CGI-I) has been widely utilized as an efficacy measure in clinical drug trials in different mental disorders.0: Very much; 1: improved; 2: Much improved; 3: Minimally improved; 4: No change; 5: Minimally worse; 6: Much worse; 7: Very much worse
Clinical global improvement scale | 1.5 years
  Clinical Global Impression Scale-improvement scale (CGI-I) has been widely utilized as an efficacy measure in clinical drug trials in different mental disorders.0: Very much; 1: improved; 2: Much improved; 3: Minimally improved; 4: No change; 5: Minimally worse; 6: Much worse; 7: Very much worse
Clinical global improvement scale | 2 years
  Clinical Global Impression Scale-improvement scale (CGI-I) has been widely utilized as an efficacy measure in clinical drug trials in different mental disorders.0: Very much; 1: improved; 2: Much improved; 3: Minimally improved; 4: No change; 5: Minimally worse; 6: Much worse; 7: Very much worse

OTHER OUTCOMES:
The symptom characteristics | 1 years
  Symptom characteristics such as tremor, type of dystonia, Parkinson's like symptoms, myoclonus, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, MD,PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol